CLINICAL TRIAL: NCT02680418
Title: A Phase I Dose Escalation Study to Assess the Pharmacokinetics (PK) of FDL169 in Healthy Female Volunteers
Brief Title: Pharmacokinetics of FDL169 in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: FDL169-2015-02
Record Dates: First submitted 2016-02-02; First posted 2016-02-11 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Single dose (Dose level 1) (Experimental): FDL169 (Dose level 1) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 2) (Experimental): FDL169 (Dose level 2) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 3) (Experimental): FDL169 (Dose level 3) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 4) (Experimental): FDL169 (Dose level 4) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 5) (Experimental): FDL169 (Dose level 5) administered as a single dose
  Interventions: Drug: FDL169
- Multiple dose (Experimental): Repeat doses of FDL169 to be administered at a dose level to be determined
  Interventions: Drug: FDL169

INTERVENTIONS:
Drug: FDL169

SUMMARY:
To determine the pharmacokinetics of single and multiple doses of FDL169 in healthy female subjects.

DETAILED DESCRIPTION:
This is a two-part study.

Part 1:

Part 1 of the study is a single-dose, dose-escalation, study to assess the safety, tolerability and PK profiles following oral administrations of FDL169 to healthy female volunteers in the fed state. Up to five doses will be assessed.

Part 2:

Part 2 of the study is a multiple-dose study to assess the safety, tolerability and PK profiles following oral administrations of FDL169 to healthy female volunteers in the fed state.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects aged 18 to 55 years inclusive and of any ethnic origin with a body mass index (BMI) of > 19 and < 30 kg/m2. Body Mass Index = Body weight (kg) / [Height (m)]
2. Subjects must be willing to use an effective method of contraception from first dose of investigational medicinal product (IMP) and for 3 months after the last dose of IMP (unless they are of non-child bearing potential).

Exclusion Criteria:

1. Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months.
2. Subjects who have any renal or clinically significant cardiac, renal or hepatic disease at Screening.
3. Subjects who have history or presence of clinically significant cardiovascular, pulmonary, renal, hepatic, haematologic, gastrointestinal (with the exception of Gilbert's syndrome or asymptomatic gallstones), endocrine or immunologic disease at Screening.
4. Have an abnormal twelve-lead ECG or an ECG with abnormality considered to be clinically significant in the opinion of the Investigator or an ECG with a single QTcB > 450 mSec.
5. Subjects with a positive urinary drugs of abuse screen or positive alcohol screen at Screening or Day -1.
6. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of > 21 units.
7. Subject with history of HIV or positive human immunodeficiency virus, hepatitis B or hepatitis C results.
8. Donation of 500 mL or more of blood within the previous 3 months.
9. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and FDL Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
10. Smoking or use of tobacco products or substitutes equivalent to > 15 cigarettes/day.
11. Any subject who is pregnant or nursing.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum plasma concentration of FDL169 (and metabolites) over 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dose
Part 1: Time to maximum plasma concentration of FDL169 (and metabolites) during 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dosing on Day 7
Part 1: Individual estimate of the terminal elimination rate constant of FDL169 (and metabolites) during 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dosing on Day 7
Part 1: Terminal half-life of FDL169 (and metabolites) during 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dosing on Day 7
Part 1: AUC from the time of dosing to the time of the last observed concentration for FDL169 (and metabolites) during 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dosing on Day 7
Part 1: AUC extrapolated to infinity from dosing time, based on the last observed concentration for FDL169 (and metabolites) during 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dosing on Day 7
Part 1: Clearance of FDL169 (and metabolites) during 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dosing on Day 7
Part 1: AUC% extrapolated for FDL169 (and metabolites) during 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dosing on Day 7
Part 2: Maximum plasma concentration of FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose
Part 2: Time to maximum plasma concentration of FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose
Part 2: Individual estimate of the terminal elimination rate constant of FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose
Part 2: Terminal half-life of FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose
Part 2: AUC from the time of dosing to the time of the last observed concentration for FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose
Part 2: AUC extrapolated to infinity from dosing time, based on the last observed concentration for FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose
Part 2: AUC from the time of dosing to time t at steady state for FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose
Part 2: Clearance of FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose
Part 2: AUC% extrapolated for FDL169 (and metabolites) following multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post-final dose) | Multiple points from pre-dose to 48 h post-final dose

SECONDARY OUTCOMES:
Number of patients with clinically significant changes in systolic blood pressure following single and multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post (final) dose) | Multiple points from pre-dose to 48 h post (last) dose
Number of patients with clinically significant changes in diastolic blood pressure following single and multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post (final) dose) | Multiple points from pre-dose to 48 h post (last) dose
Number of patients with clinically significant changes in pulse rate following single and multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post (final) dose) | Multiple points from pre-dose to 48 h post (last) dose
Number of patients with clinically significant changes in oxygen saturation following single and multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post (final) dose) | Multiple points from pre-dose to 48 h post (last) dose
Number of patients with clinically significant changes in oral temperature following single and multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post (final) dose) | Multiple points from pre-dose to 48 h post (last) dose
Number of patients with clinically significant 12-lead ECG abnormalities following single and multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post (final) dose) | Multiple points from pre-dose to 48 h post (last) dose
Number of patients with abnormal laboratory values following single and multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post (final) dose) | Multiple points from pre-dose to 48 h post (last) dose
Number of patients experiencing treatment-related adverse events following single and multiple oral doses of FDL169 (assessed throughout dosing and for 48 h post (final) dose) | Multiple points from pre-dose to 48 h post (last) dose

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abou-Farha, MBChB MD PhD, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, Wales, United Kingdom